CLINICAL TRIAL: NCT00439907
Title: A Prospective, Randomized Study Comparing the Outcome of Overlap and End-to-end Repair in Anal Sphincter Rupture During Delivery
Brief Title: Comparison of Overlap and End-to-end Repair in Anal Sphincter Rupture During Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SF2005-07
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2010-08

CONDITIONS: Rupture; Childbirth
Keywords: Anal sphincter Delivery; Primary repair; End-to-end repair; Over-lap repair; Anal manometry; Anal sonography; Weksner Score; Rupture of the external anal sphincter during delivery; Anal sphincter; Anal sphincter rupture
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- End-to-end (Active Comparator): End-to-end repair
  Interventions: Procedure: End-to-end repair of the external anal sphincter muscle
- Overlap (Active Comparator): Overlap repair
  Interventions: Procedure: Overlap repair of the external anal sphincter muscle

INTERVENTIONS:
Procedure: End-to-end repair of the external anal sphincter muscle — Surgical procedure: End-to-end repair of the external anal sphincter muscle
  Arms: End-to-end
Procedure: Overlap repair of the external anal sphincter muscle — Surgical procedure: Overlap repair of the external anal sphincter muscle
  Arms: Overlap

SUMMARY:
Rupture of the external anal sphincter occurs in about 4% percent of deliveries. It is not clear from other studies whether the results concerning anal function, e.g. fecal continence, are better with the overlap repair or end-to-end repair of the injured muscle. The researchers randomize women at birth to either overlap or end-to-end when the injury is recognized, and examine them one year later with special anal physiologic examinations and a validated questionnaire. The hypothesis is that the overlap technique is superior.

DETAILED DESCRIPTION:
Rupture of the external anal sphincter occurs in about 4% percent of deliveries in our department. It is not clear from other studies whether the results concerning anal function are better with the overlap repair or end-to-end repair of the injured muscle. Our routine has been to perform an end-to-end repair, though anal surgeons, in the setting of a secondary repair, prefer the overlap method. Former studies, when the repair was performed by highly skilled operators, have indicated that the overlap method is better.

We wanted to compare the two methods through a RCT with the end-points examination results after one year addressing endoanal sonography findings, anal manometric results and continence score evaluated by a Weksner score questionnaire. Our study is performed in the routine clinical setting. The patients are recruited to the study during delivery when the injury is recognized. When she has given her informed consent she is randomized to one of the two operation methods. The operation is performed by the consultant obstetrician on call or the resident supervised by the consultant. The proctologist who performs the anal manometry and sonography after one year is blinded to the surgical method.

We plan to include approximately 160 patients at one center. In our center we have about 4500 deliveries per year.

ELIGIBILITY:
Inclusion Criteria:

* Delivery
* Anal sphincter rupture

Exclusion Criteria:

* Lack of ability to understand the informed consent form
* Lack of ability to cooperate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-02; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Anal Sonography | pre-partum
Endoanal manometry | pre-partum

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Rygh, MD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Background] Sultan AH, Monga AK, Kumar D, Stanton SL. Primary repair of obstetric anal sphincter rupture using the overlap technique. Br J Obstet Gynaecol. 1999 Apr;106(4):318-23. doi: 10.1111/j.1471-0528.1999.tb08268.x. PMID 10426237
- [Background] Fitzpatrick M, Behan M, O'Connell PR, O'Herlihy C. A randomized clinical trial comparing primary overlap with approximation repair of third-degree obstetric tears. Am J Obstet Gynecol. 2000 Nov;183(5):1220-4. doi: 10.1067/mob.2000.108880. PMID 11084569
- [Derived] Rygh AB, Korner H. The overlap technique versus end-to-end approximation technique for primary repair of obstetric anal sphincter rupture: a randomized controlled study. Acta Obstet Gynecol Scand. 2010 Oct;89(10):1256-62. doi: 10.3109/00016349.2010.512073. PMID 20846058